CLINICAL TRIAL: NCT05650996
Title: The Impact of Early ADL Participation on Functional Outcomes Post Distal Radius Fracture
Brief Title: Impact of Early ADL Participation on Outcomes Post DRF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: American Hand Therapy Foundation (Unknown)
Responsible Party: Principal Investigator, Sarah Doerrer, Assistant Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCR224559
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Distal Radius Fracture
Keywords: Activities of Daily Living; Patient Education
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADL video/Cast Care (Experimental): ADL/cast care instructional video ADL/cast care handout
  Interventions: Behavioral: ADL/Cast Care instruction; Behavioral: Cast Care Instruction
- Cast Care Video (Active Comparator): Cast care instructional video Cast care handout
  Interventions: Behavioral: Cast Care Instruction

INTERVENTIONS:
Behavioral: ADL/Cast Care instruction — Participants in the experimental group will watch a video instructing them on early ADL participation after DRF fracture treated in a cast and cast care. Participants in the experimental group will also receive a handout on ADL participation and cast care.
  Arms: ADL video/Cast Care
Behavioral: Cast Care Instruction — Participants in the control group will watch a video instructing them on cast care. Participants in the control group will receive a handout on cast care.

SUMMARY:
This study is a randomized controlled trial (RCT). This RCT which will study the effect of performing daily activities early after a distal radius fracture being treated conservatively in a cast. This study will have two groups. The experimental group will watch a video and be given a handout on how to perform daily activities with the hand of the injured wrist while in a cast and cast care. The control group will watch a video on cast care and be given a handout on cast care. Outcome measures will be taken at initial evaluation between 0-3 weeks, at 6 weeks, at 9 weeks, and at 3 months. Outcome measures will include the Michigan Wrist Evaluation, Visual Analog Pain Scale, Tampa Scale of Kinesiophobia-11 Scale, finger mobility testing, grip and pinch strength, and the 9 hole peg test to test fine motor coordination. Outcome measure scores will be compared between groups using a t-test statistical test. Outcome measure scores will also be tested within groups using a paired t-test.

DETAILED DESCRIPTION:
1. The surgeon will recruit patients who have met inclusion and exclusion criteria utilizing a recruitment statement.
2. If the patient is interested in participating in the study, the surgeon will obtain informed consent and email a copy of the informed consent form to the patient.
3. Once informed consent is obtained, the surgeon will ask the front desk to give him an envelop which will include a letter with either the word control or experimental group on it. Once the surgeon reads the letter, the subject will receive either the standard of care video and handout (control) or the intervention video and handout (experimental).
4. If the subject receives the intervention then the surgeon will play the intervention video in the office and review with the subject the educational handout. The handout will be given to the subject to take home and a link to the handout and video will be emailed to the subject.
5. If the subject is in the control group then the surgeon will play the standard of care (cast care) video in the office and review with the subject the cast care handout. The handout will be given to the subject to take home and a link to the handout and video will be emailed to the subject.

The following data collection procedures will occur with the subjects

The surgeon will collect data from all subjects at 0-3 weeks post injury and data collection will include: age, gender, race, hand dominance, side injured, fracture severity, workers comp status, comorbidities, smoker status, work status, and household assistance. The hand surgeon will also collect data from the subjects on their current level of function, pain, and fear of moving their injured limb.

At 6 weeks the surgeon will collect data from all subjects on their current level of function, pain, fear of moving their injured limb. The surgeon will also measure finger motion.

At 9 weeks the surgeon will collect data from all subjects on their current level of function, pain, fear of moving their injured limb. The surgeon will also measure finger motion, grip, pinch strength and fine motor coordination.

At 3 months the surgeon will collect data from all subjects on their current level of function, pain, fear of moving their injured limb. The surgeon will also measure finger motion, grip, pinch strength and fine motor coordination.

All subjects will be followed for 3 months. If at 6 weeks or later the patient receives a referral for hand therapy it will be noted in the record. It will also be noted in the record if subject experiences any complication such as median nerve compression, tendonitis, or complex regional pain syndrome.

The outcome measures that will be used with both the control and experimental groups and at each time point that the data will be collected. All outcome measures will be uploaded onto RedCap. Subjects will use a tablet to fill out all questionnaires (Michigan Hand Evaluation, Visual Analog Scale, Tampa Scale of Kinesiophobia-11) while in the office or forms will be emailed through RedCap and scores will be uploaded into the RedCap database. All clinical tests (grip and pinch testing, distance from distal palmar crease, 9 hole peg test) will be recorded in RedCap. Demographic information will either be collected on the tablet in RedCap.

ELIGIBILITY:
Inclusion Criteria:

English Speaking

DRFs treated with a cast

Individuals over the age of 18

Less than 3 weeks from DRF

Exclusion Criteria:

Individuals with pre-existing neurological conditions affecting the upper limb

Individuals with cognitive deficits that would limit the ability to correctly report information on outcome measures

Individuals with psychological deficits which would limit the ability to correctly report information on outcome measures

Individuals with multiple injuries to the affected upper limb

Individuals with multiple injuries to both upper limbs

Individuals requiring surgery to fixate the distal radius fracture

Prior distal radius fracture involving the same wrist

Individuals receiving hand therapy for another injury at enrollment into study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Michigan Hand Questionnaire | baseline
  Patient reported outcome measure for function, min value-0 max value-100 , higher score is best possible ability
Michigan Hand Questionnaire | 6 weeks
  Patient reported outcome measure for function, min value-0 max value-100 , higher score is best possible ability
Michigan Hand Questionnaire | 9 weeks
  Patient reported outcome measure for function, min value-0 max value-100 , higher score is best possible ability
Michigan Hand Questionnaire | 3 months
  Patient reported outcome measure for function, min value-0 max value-100 , higher score is best possible ability
Visual Analog Scale | baseline
  patient reported outcome measure for pain intensity, max value=100, min value=0, higher score is more pain
Visual Analog Scale | 6 weeks
  patient reported outcome measure for pain intensity, max value=100, min value=0, higher score is more pain
Visual Analog Scale | 9 weeks
  patient reported outcome measure for pain intensity, max value=100, min value=0, higher score is more pain
Visual Analog Scale | 3 months
  patient reported outcome measure for pain intensity, max value=100, min value=0, higher score is more pain
Tampa Scale of Kinesiophobia | baseline
  patient reported outcome measure for fear of movement, min score=11 max score=44, higher score indicates more kinesiophobia
Tampa Scale of Kinesiophobia | 6 weeks
  patient reported outcome measure for fear of movement, min score=11 max score=44, higher score indicates more kinesiophobia
Tampa Scale of Kinesiophobia | 9 weeks
  patient reported outcome measure for fear of movement, min score=11 max score=44, higher score indicates more kinesiophobia
Tampa Scale of Kinesiophobia | 3 months
  patient reported outcome measure for fear of movement, min score=11 max score=44, higher score indicates more kinesiophobia
Range of motion of digits | 6 weeks
  distance from digits to distal palmar crease, min score=0, score of 0 signifies that the individual can touch the palm
Range of motion of digits | 9 weeks
  distance from digits to distal palmar crease, min score=0, score of 0 signifies that the individual can touch the palm
Range of motion of digits | 3 months
  distance from digits to distal palmar crease, min score=0, score of 0 signifies that the individual can touch the palm
Grip and Pinch Strength | 9 weeks
  Jamar grip gauge testing and pinchmeter gauge testing for strength. Min score=0, higher score indicates more strength
Grip and Pinch Strength | 3 months
  Jamar grip gauge testing and pinchmeter gauge testing for strength. Min score=0, higher score indicates more strength
9 hole peg test | 9 weeks
  fine motor coordination/sensorimotor test. Timed test therefore a longer time to complete reflects reduced finger dexterity
9 hole peg test | 3 months
  fine motor coordination/sensorimotor test. Timed test therefore a longer time to complete reflects reduced finger dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Facilities Associates, Washington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No